CLINICAL TRIAL: NCT02230150
Title: ADHESION TO THERAPEUTIC STRATEGIES FOR OUTPATIENTS WITH HEART FAILURE - ADhesion-HF
Acronym: ADhesion-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Márcia Maria Carneiro Oliveira, ADHESION TO THERAPEUTIC STRATEGIES FOR OUTPATIENTS WITH HEART FAILURE, Federal University of Bahia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ADhesion-HF
Record Dates: First submitted 2014-08-20; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure
Keywords: Adhesion, Knowledge, Nursing
MeSH Terms: conditions — Heart Failure; Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Adhesion-HF — The hypothesis that was investigated is whether the nursing consultation improves therapeutic strategies for membership, adherence to self-care, improved levels of NT-proBNP improves performance in 6-minute walk test, monitoring of biomarkers of laboratory tests (sodium , potassium, urea, creatinine and NT-proBNP) frequent occurrence of readmissions and mortality in patients with heart failure after 1 month.

SUMMARY:
The purpose of this study is to verify the impact of the educational intervention in the adhesion to therapeutic strategies for patients with heart failure.

DETAILED DESCRIPTION:
1. Characterize the socio-demographic and clinical aspects of heart failure patients;
2. Awareness before and after nursing consultation, in relation to diet for heart failure, liquid and weight, general heart failure information, medication, physical activity, measures to improve disease control, signs of decompensated heart failure;
3. Adhesion of patients before and after nursing consultation, related to medication, liquid and weight, use of alcohol and importance of returning for consultation and exams.
4. Evaluated the impact of educational intervention at the levels of NT-proBNP, urea, creatinine, sodium, potassium, before and after nursing consultation;
5. The 6 minute walk test performance before and after nursing consultation;
6. The distance covered and time of the 6 minute walk test, until fatigue in heart failure patients before and after nursing consultation;

ELIGIBILITY:
Inclusion Criteria:

* During the first phase of the study all the heart failure patients with ventricular ejection fraction of up to 49% shall be included (confirmed through ECOTT performed during the past year). All patients inserted had systolic heart failure and were scheduled and which agreed to take part of the research, signing a term of informed consent.

Exclusion Criteria:

* Individuals with cognitive deficit, first outpatient medical consultation, suffered AMI (acute myocardial infarction) within the last 3 months or a stroke, post-operative of cardiac surgery, patients with chronic obstructive pulmonary disease (COPD), orthopedic problems, patients over the age of 80 and those that do not accept to participate of the research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
ADHESION TO THERAPEUTIC STRATEGIES FOR OUTPATIENTS WITH HEART FAILURE | 1 month
  Verify the impact of the educational intervention in the adhesion to therapeutic strategies for patients with heart failure.

SECONDARY OUTCOMES:
changes in biomarkers: Nt-proBNP, sodium, potassium, urea and creatinine | 1 month
  changes in biomarkers: Nt-proBNP, sodium, potassium, urea and creatinine before and after nursing consultation

OTHER OUTCOMES:
performance in the six minutes walk test | 1 month
  monitor the difference in performance of the 6-minute walk test in adherent and non-adherent

CONTACTS AND LOCATIONS:
Overall Officials: Márcia M Carneiro Oliveira, Principal Investigator
Locations (1):
- Hospital Ana Nery, Salvador, Estado de Bahia, Brazil